CLINICAL TRIAL: NCT02960399
Title: Assessment of Immunogenicity of Zostavax® in Patients With Antibody Deficiency 60 Years of Age and Older
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI has terminated the study at this time.
Sponsor: University of South Florida (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00023706
Record Dates: First submitted 2016-10-03; First posted 2016-11-09 (Estimated); Last update posted 2018-05-31 (Actual); Status verified 2018-04

CONDITIONS: Common Variable Immune Deficiency; Specific Antibody Deficiency; X-linked Agammaglobulinemia
MeSH Terms: conditions — Common Variable Immunodeficiency; Bruton type agammaglobulinemia | interventions — Herpes Zoster Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Antibody Deficient Patients (Experimental): Zostavax® vaccine administered to antibody deficient patients 60 years of age and older.
  Interventions: Biological: Zostavax®
- Healthy Subjects (Active Comparator): Zostavax® vaccine administered per standard of care to healthy adults 60 years of age and older.
  Interventions: Biological: Zostavax®

INTERVENTIONS:
Biological: Zostavax® — Zostavax® immunization

SUMMARY:
Recommendations concerning the administration of Zostavax® in patients with antibody deficiency are unclear. The investigators plan to assess the immunogenicity and safety of Zostavax® in patients with antibody deficiency as compared with healthy volunteers.

DETAILED DESCRIPTION:
Common variable immune deficiency (CVID), specific antibody deficiency (SAD), and X-linked agammaglobulinemia (XLA) are among the most common primary antibody deficiencies in which the mainstay of treatment is gammaglobulin replacement. The use of high doses of immunoglobulin replacement therapy and the early recognition of co-morbid diseases during the course of CVID, SAD, and XLA has improved survival and led to an aging population of CVID, SAD, and XLA patients.

The Advisory Committee on Immunization Practices (ACIP) recommends routine vaccination of all persons aged >60 years with 1 dose of vaccine directed against herpes zoster (Zostavax®) in the absence of any contraindications. Current standard of care includes avoidance of all vaccines when receiving gammaglobulin products due to passive immunity obtained from gammaglobulin against vaccine preventable infections. The exception to this rule is that patients on gammaglobulin should receive the yearly influenza vaccine due to its enhanced cell mediated immunity against the influenza virus. Clinical immunologists currently have no data upon which to advise patients receiving gammaglobulin replacement including those with CVID, SAD, and XLA concerning use of Zostavax®.

All gammaglobulin replacement products maintain protective antibody levels against VZV. However, humoral immune responses with anti-VZV antibodies are relatively constant and do not protect against the development of shingles. Varicella zoster virus specific cell mediated immunity (VZV-CMI), which is T cell dependent, is the critical component in preventing herpes zoster (shingles). VZV-CMI diminishes with age leaving the elderly most susceptible to shingles. Several studies have concluded that boosting VZV-CMI protects older adults from developing herpes zoster and postherpetic neuralgia (PHN).

Recommendations on the prevention of herpes zoster published in the Morbidity and Mortality Weekly Report (MMWR) by the Centers for disease control (CDC) in May 2008 make the following statements:

1. Zoster vaccine should not be administered to persons with primary or acquired immunodeficiency including:

   a. Persons with clinical or laboratory evidence of other unspecified cellular immunodeficiency.
2. Persons with impaired humoral immunity (e.g., hypogammaglobulinemia or dysgammaglobulinemia) can/should receive zoster vaccine.

The investigators hypothesize that vaccination with Zostavax® in adults with CVID, SAD, and XLA who have evidence of normal cell mediated immunity with normal T cell quantities and function will have a boost in VZV-CMI thereby reducing susceptibility to shingles and PHN.

Successful completion of this study will provide clinical immunologists with data upon which to advise antibody deficient patients concerning the use of Zostavax®.

ELIGIBILITY:
Inclusion/Exclusion Criteria for Antibody Deficient Patients

Inclusion Criteria

* Adults 60 years of age and older
* Diagnosis of common variable immunodeficiency (CVID), Specific Antibody Deficiency (SAD), or X-linked agammaglobulinemia (XLA)
* Receiving replacement gammaglobulin
* Willing and able to sign consent and follow study schedule
* History of varicella or long-term (greater than or equal to 30 years) residence in the USA

Exclusion Criteria

* Allergy to Zostavax® or any of its components (i.e gelatin, neomycin)
* Absolute CD3, CD4, or CD8 lymphopenia as determined by age specific reference ranges
* Poor T cell function as indicated by a < 30 % increase in T cell response to mitogens or antigens as compared to the age matched normal reference range (in CVID) subjects
* Evidence of acute systemic illness or infection at within four weeks of screening or enrollment
* Prior herpes zoster infection
* Previously received herpes zoster vaccination
* Malignancy including solid tumors, leukemia, or lymphoma
* Presence of autoimmune or other inflammatory disease
* Use of immunosuppressive or immunomodulatory medications including chronic corticosteroids. Treatment for >2weeks of daily steroids will be considered chronic use.
* History of bleeding or chronic skin disorders.
* Pregnant or breastfeeding females
* Immunizations within one month
* Persons with HIV or AIDS
* Subject unwilling to sign consent or adhere to study schedule
* Any condition that in the opinion of the investigator would interfere with the conduct of the study
* Subjects unlikely to adhere to protocol follow-up

Inclusion/Exclusion Criteria for Healthy Subjects

Inclusion Criteria

* Adults 60 years of age and older
* Willing and able to sign consent and follow study schedule
* History of varicella or long-term (greater than or equal to 30 years) residence in the USA

Exclusion Criteria

* Allergy to Zostavax® or any of its components (i.e gelatin, neomycin)
* Evidence of acute systemic illness or infection at within four weeks of screening or enrollment
* Prior herpes zoster infection
* Previously received herpes zoster vaccination
* Malignancy including solid tumors, leukemia, or lymphoma
* Presence of autoimmune or other inflammatory disease
* Use of immunosuppressive or immunomodulatory medications including chronic corticosteroids. Treatment for >2weeks of daily steroids will be considered chronic use.
* History of bleeding or chronic skin disorders.
* Pregnant or breastfeeding females
* Immunizations within one month
* Persons with HIV or AIDS
* Subject unwilling to sign consent or adhere to study schedule
* Any condition that in the opinion of the investigator would interfere with the conduct of the study
* Subjects unlikely to adhere to protocol follow-up

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-12; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Determine in vitro changes in T cell proliferation preceding and following vaccination with Zostavax® by measurement of lymphocyte proliferation in response to VZV antigen. | Day 0, Week 4, 3 months, 6 months
  Determine in vitro lymphocyte proliferation as counts per minute after stimulation of cells with varicella zoster antigen at time points preceding and following vaccination with Zostavax. Blood samples will be obtained prior to administering the Zostavax® vaccine and post-vaccination at 4 weeks, 3 months, and 6 months.

SECONDARY OUTCOMES:
Determine in vitro changes in T cell proliferation preceding and following vaccination with Zostavax® by measurement of IFNg production by T cells in response to VZV antigen. | Day 0, Week 4, 3 months, 6 months
  Determine in vitro IFNg production as Units/ml after stimulation of cells with varicella zoster antigen at time points preceding and following vaccination with Zostavax. Blood samples will be obtained prior to administering the Zostavax® vaccine and post-vaccination at 4 weeks, 3 months, and 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Leiding, MD, Principal Investigator — University of South Florida
Locations (1):
- University of South Florida, St. Petersburg, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided